CLINICAL TRIAL: NCT07361926
Title: Sexual Health Access at Retail Pharmacies: Advancing Pharmacy-based Delivery of Primary STI and HIV Prevention for Cisgender Women
Acronym: SHARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jillian Pintye, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022204; R01HD118713 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sexually Transmitted Infections (Not HIV or Hepatitis); HIV Infections
Keywords: STI prevention; HIV prevention; Pharmacy delivery
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis; HIV Infections | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: 3 arm, non blinded, individually randomized controlled trial to compare 1) HIV PEP/PrEP plus serial STI testing and non doxy-PEP, 2) HIV PEP/PrEP plus serial STI testing alone, and 3) HIV PEP/PrEP only, with embedded mixed-methods implementation and economic evaluation components.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Serial STI testing and doxy-PEP (Active Comparator): STI testing and doxy-PEP offered with HIV PEP/PrEP services
  Interventions: Drug: doxy-PEP; Diagnostic Test: Serial STI testing; Drug: HIV PEP/PrEP
- Serial STI testing alone (Active Comparator): STI testing offered with HIV PEP/PrEP
  Interventions: Diagnostic Test: Serial STI testing; Drug: HIV PEP/PrEP
- No serial STI testing or doxy-PEP (Active Comparator): HIV PEP/PrEP services only
  Interventions: Drug: HIV PEP/PrEP

INTERVENTIONS:
Drug: doxy-PEP — Antiobiotic for post exposure prophylaxis
  Other Names: doxycycline
  Arms: Serial STI testing and doxy-PEP
Diagnostic Test: Serial STI testing — CT/NG and syphilis testing
  Arms: Serial STI testing alone; Serial STI testing and doxy-PEP
Drug: HIV PEP/PrEP — HIV post and pre exposure prophylaxis

SUMMARY:
This proposed 3-arm randomized study will compare different pharmacy based approaches that include HIV prevention medication (PrEP and PEP), routine STI testing, and preventive antibiotic (doxycycline) for STIs. The study will assess how well these services can be implemented, how acceptable they are to young women, and whether they are cost-effective.

DETAILED DESCRIPTION:
Global incidence of STIs increased over the past decade, with over one million curable STIs acquired daily. In 2020, the World Health Organization (WHO) estimated 374 million new infections of Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), Trichomonas vaginalis (TV), and syphilis. Young women in East Africa face high prevalence of curable STIs and HIV,4 and high STI incidence. Studies confirm higher STI prevalence among younger women compared to their male peers, and older women. STIs severely affect mortality and morbidity for cisgender women by causing tubal infertility, chronic pelvic pain, pelvic inflammatory disease, ectopic pregnancy, postpartum endometriosis, adverse neonatal outcomes, and increased susceptibility to HIV. In HIV high-burden settings, cultural, economic, and social marginalization of women contributes to the risk of HIV and STIs,10 in part by making condom use negotiation challenging. Despite high STI burden in these settings, research to address STIs lags behind HIV in young cisgender women.

WHO calls for vastly increasing STI testing and integrating STI interventions to reach priority populations.Sexually transmitted infections (STIs) disproportionately affect cisgender adolescent girls and young women (AGYW) who often experience STI complications, including infertility, chronic pelvic pain, and increased risk for HIV acquisition and peripartum morbidity. In Kenya, HIV and STIs comprise a syndemic with 40% of new HIV infections occurring among AGYW. Yet, research to address STIs lags behind HIV in this priority population and no primary STI prevention tools are currently available to cisgender women beyond condoms. In Kenya, 40% of women access contraception without interfacing with facilities, including at retail pharmacies, and are missed by facility-based HIV services like pre-exposure prophylaxis (PrEP). In the ongoing work among AGYW seeking contraception at 20 pharmacies in Kisumu, Kenya (NCT05467306); all AGYW offered STI testing accepted, 29% had CT or NG, and 70% accepted expedited partner therapy (EPT) and report no social harms. Among AGYW seeking emergency contraception, only 3% previously used HIV post-exposure prophylaxis (PEP), highlighting an opportunity to offer HIV PEP to AGYW via pharmacies. Qualitative data suggest that STI testing motivates health promoting behaviors, even when STI results are negative.

To date, no studies evaluate if serial STI testing promotes PrEP persistence. 'Event-driven' doxycycline PEP (doxy-PEP) for CT, NG, and syphilis found no protective benefit for Kenyan women accessing PrEP at facilities, likely due to low adherence. AGYW more frequently access emergency contraception at pharmacies compared to facilities; thus, 'event-driven' strategies, like HIV PEP ("PEP-in-Pocket") or doxy-PEP, may have higher use in pharmacies. The investigators propose a RCT in Kisumu, Kenya-a region with 11% HIV prevalence-to test co-offering HIV PEP/PrEP and STI testing with and without doxy-PEP in pharmacies and prospectively assess HIV PEP/PrEP use and persistence, and STI incidence among AGYW (n=720) and estimate cost and cost-effectiveness of this strategy. The investigators hypothesize that expanding HIV and STI prevention options to include HIV PEP, STI testing, EPT, and doxy-PEP in pharmacies will be cost-effective and improve HIV and STI outcomes in AGYW, a population disproportionately affected by STIs and HIV. The study is designed to inform pharmacy delivery of biomedical HIV and STI prevention services and provide evidence to inform policy for STI/HIV prevention among AGYW.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender female
* Seeking contraception (emergency contraception, oral contraceptive pills, injectables, implants, and condoms) from the retail pharmacy site
* Age ≥ 15 and <25 years old
* Willingness to receive PrEP screening per national guidelines including HIV testing
* Not currently taking PrEP
* Planning to reside in the area for the next 12 months
* Able and willing to provide informed consent for participation

Exclusion Criteria:

* Current participation in other ongoing studies.
* Medical contraindications to PrEP or doxycycline use (e.g., severe allergy to doxycycline, serious hepatic or renal disease).
* Any other condition that, in the investigator's judgment, would make participation unsafe or interfere with study procedures.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cis-gender female
Enrollment: 720 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
HIV PrEP initiation | From enrollment to the end of participant follow up after 12 months
  HIV PrEP initiation among women seeking contraception at retail pharmacies defined as accepting either daily oral PrEP pills or the DPV-VR when offered at enrollment and evidence of self-reported use at 1-month post-acceptance
HIV PrEP persistence | From enrollment to the end of participant follow up at 12 months
  PrEP persistence defined as continuing with HIV PrEP use at 12-months
STI incidence | From enrollment to the end of participant follow up at 12 months
  STI incidence (CT, NG, and/or syphilis)

SECONDARY OUTCOMES:
HIV PEP, PrEP method selection | From enrollment to the end of participant follow up at 12 months
  Self-selection of DPV-VR, daily PrEP, and/or PEP when offered at enrollment compared across all randomization arms
HIV PrEP following PEP | From enrollment to the end of participant follow up at 12 months
  Initiating HIV PrEP at anytime of the study following prior HIV PEP use
HIV PrEP adherence | At end of participant follow up at 12 months
  Detectable TFC levels in hair at 12 month visit
Predictors of non-adherence | From enrollment through the end of participant follow up at 12 months
  Factors associated with poor adherence (<90% adherence on PrEP or discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Pintye, PhD, Principal Investigator — University of Washington